CLINICAL TRIAL: NCT03329378
Title: A Phase II Randomized Trial Evaluating Neoadjuvant Dose-Dense Doxorubicin/Cyclophosphamide Followed by Paclitaxel/Trastuzumab/Pertuzumab (AC THP) and Docetaxel/Carboplatin/Trastuzumab/Pertuzumab (TCHP) For Early Her2Neu Positive Breast Cancer
Brief Title: Neoadjuvant Dose-Dense For Early Her2Neu Positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data Safety Monitoring Board is in agreement with the study findings so far and the stopping rule has been met, which suspends the study treatment arms in March 2021.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Aarti S. Bhardwaj, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-1585
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Locally Advanced Breast Cancer
Keywords: Neoadjuvant chemotherapy; locally advanced breast cancer; Her2neu
MeSH Terms: interventions — Docetaxel; Carboplatin; Trastuzumab; pertuzumab; pegfilgrastim; Paclitaxel; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ddACTHP (Active Comparator): Doxorubicin 60 mg/m2 IV day 1 Cyclophosphamide 600 mg/m2 IV day 1 Pegfilgrastim 6mg SC, day 2 of AC
  Cycled every 14 days for 4 cycles, followed by, Paclitaxel 80 mg/m2 IV x 1 hour infusion on days 1, 8, and 15 Trastuzumab 8 mg/kg IV day 1, followed by 6mg/kg Pertuzumab loading dose 840 mg IV followed by 420 mg IV every 3 weeks
  Cycled every 21 days for 4 cycles, followed by, Trastuzumab 6mg/kg every 21 days to complete 1 year
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide
- TCHP (Active Comparator): TCHP (Docetaxel, Carboplatin, Trastuzumab, Pertuzumab, Pegfilgrastim ) institutional practice is to titrate the infusion rate on the initial Paclitaxel dose (40 ml/hr x 5 min, then 80 ml/hr x 5 min, then 120 ml/hr x 10 min, then 200 ml/hr). Subsequent Paclitaxel doses are given over 1 hour.
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Pegfilgrastim; Drug: Paclitaxel

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75mg/m2 IV, day 1
  Arms: TCHP
Drug: Carboplatin — Carboplatin AUC 6 IV, day 1
  Arms: TCHP
Drug: Trastuzumab — Trastuzumab 8mg/kg IV initial dose, followed by 6mg/kg IV , day 1
  Arms: TCHP
Drug: Pertuzumab — Pertuzumab 840 mg IV initial dose followed by 420 mg IV, day 1
Drug: Pegfilgrastim — Pegfilgrastim 6mg SC, day 2 Cycled as per arm
  Arms: TCHP
Drug: Trastuzumab — Trastuzumab 6mg/kg every 21 days to complete 1 year
Drug: Paclitaxel — Titrate the infusion rate on the initial Paclitaxel dose (40 ml/hr x 5 min, then 80 ml/hr x 5 min, then 120 ml/hr x 10 min, then 200 ml/hr). Subsequent Paclitaxel doses are given over 1 hour.
Drug: Doxorubicin — Doxorubicin 60 mg/m2 IV day 1
  Arms: ddACTHP
Drug: Cyclophosphamide — Cyclophosphamide 600 mg/m2 IV day 1
  Arms: ddACTHP
Drug: Paclitaxel — 80 mg/m2 IV x 1 hour infusion on days 1, 8, and 15
  Arms: ddACTHP

SUMMARY:
Primary Objective:

• Determination of pathologic complete response (pCR) rates

Secondary Objective:

* Determination of cardiac toxicity as measured by: composite of LVEF, longitudinal strain and troponin.
* Breast conservation rates
* Overall survival

Study Design

* Approximately 34-74 patients with Her2 positive, Stage II-regional IV breast cancer will be enrolled.
* Patients will be stratified by ER/PR status.
* They will be randomized to ddACTHP vs TCHP.

  * Initially, 17 patients will be randomly assigned to each treatment arm.
  * If 3 or fewer patients have a pCR, then that arm will be terminated and no further patients will be entered on that treatment arm.
  * If 4 or more patients obtain a pCR, 20 additional patients (total of 37 patients) will be randomized to that treatment arm.
  * If 11 or more patients out of 37 have a pCR, the treatment will be of interest for further study.

ELIGIBILITY:
Inclusion Criteria:

The patient must have signed and dated an IRB-approved consent form that conforms to federal and institutional guidelines.

* Female
* 18 years or older
* ECOG performance status of 0 or 1
* Eligible tumors must meet one of the following criteria:

  * Operable (T1c, T2-3, N0-1, M0)
  * Locally advanced (T2-3, N2-3, M0 or T4a-c, any N, M0)
  * Inflammatory breast cancer (T4d, any N, M0)
* Staging evaluation:

  * History and physical exam, cbc, chemistry profile
  * CT Chest/Abdomen/Pelvis and a bone scan or PET/CT as needed
* Diagnosis of invasive adenocarcinoma made by core needle biopsy
* Breast cancer determined to be:
* Confirmed HER2-positive : (ASCO CAP guidelines, 10/7/2013)

  * IHC 3+ based on circumferential membrane staining that is complete, intense
  * ISH positive based on:
  * Single probe average HER2 copy number ≥ 6 signals/cell
  * Dual probe HER2/CEP 17 ratio ≥ 2.0 with an average HER2 copy number ≥ 4.0 signals/cell
  * Dual probe HER2/CEP 17 ratio ≥ 2.0, with an average HER2 copy number of < 4.0 signals/cell
  * Dual probe HER2/CEP 17 ratio < 2.0 with the average HER2 copy number of ≥ 6.0 signals/cell
* any ER or PR receptor status
* LVEF assessment by echocardiogram within 30 days of initiation; EF of ≥ 55% considered normal.
* Normal troponin I level at baseline
* Blood counts must meet the following criteria:

  * ANC greater than or equal to 1500/mm3
  * Platelet count greater than or equal to 100,000/mm3
  * Hemoglobin greater than or equal to 10 g/dL
* Serum creatinine less than or equal 2.5 mg/100ml
* Adequate hepatic function by these criteria: total bilirubin must be less than or equal to 1.5 x the ULN for the lab unless the patient has a bilirubin elevation great than the ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and alkaline phosphatase must be less than or equal to 2.5 x ULN for the lab; and AST must be less than or equal to 1.5 x ULN for the lab. Both alkaline phosphatase and AST may not both be greater than the ULN.
* Patients with AST or alkaline phosphatase > ULN are eligible for inclusion in the study if liver imaging (CT, MRI, PET-CT or PET scan) performed within 90 days prior to randomization does not demonstrate metastatic disease and the requirements are met as above
* Patients with alkaline phosphatase that is > ULN but less than or equal to 2.5 x ULN or unexplained bone pain are eligible for inclusion in the study if a bone scan, PET-CT scan, or PET scan performed within 90 days prior to randomization does not demonstrate metastatic disease.

Exclusion Criteria:

Patients with a history of decompensated congestive heart failure or an EF < 55% will be excluded

• Cardiac disease that would preclude the use of the drugs included in the above regimens. This includes but is not confined to:

* Active cardiac disease:
* angina pectoris requiring the use of anti-anginal medication;
* ventricular arrhythmias except for benign premature ventricular contractions controlled by medication;
* conduction abnormality requiring a pacemaker;
* supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication; and
* clinically significant valvular disease
* symptomatic pericarditis
* pulmonary hypertension
* History of cardiac disease:
* myocardial infarction;
* congestive heart failure; or
* cardiomyopathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2021-03-07 (Actual); Study Completion 2021-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aarti Bhardwaj, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Mount Sinai Beth Israel, New York, New York
  - Mount Sinai West, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ddACTHP: Doxorubicin 60 mg/m2 IV day 1 Cyclophosphamide 600 mg/m2 IV day 1 Pegfilgrastim 6mg SC, day 2 of AC
  Cycled every 14 days for 4 cycles, followed by, Paclitaxel 80 mg/m2 IV x 1 hour infusion on days 1, 8, and 15 Trastuzumab 8 mg/kg IV day 1, followed by 6mg/kg Pertuzumab loading dose 840 mg IV followed by 420 mg IV every 3 weeks
  Cycled every 21 days for 4 cycles, followed by, Trastuzumab 6mg/kg every 21 days to complete 1 year
  Pertuzumab: Pertuzumab 840 mg IV initial dose followed by 420 mg IV, day 1
  Trastuzumab: Trastuzumab 6mg/kg every 21 days to complete 1 year
  Paclitaxel: Titrate the infusion rate on the initial Paclitaxel dose (40 ml/hr x 5 min, then 80 ml/hr x 5 min, then 120 ml/hr x 10 min, then 200 ml/hr). Subsequent Paclitaxel doses are given over 1 hour.
  Doxorubicin: Doxorubicin 60 mg/m2 IV day 1
  Cyclophosphamide: Cyclophosphamide 600 mg/m2 IV day 1
  Paclitaxel: 80 mg/m2 IV x 1 hour infusion on days 1, 8, and 15
Period: Overall Study
Arm/Group | ddACTHP | TCHP
Started | 2 | 5
Completed | 2 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ddACTHP | TCHP | Total
Number analyzed (Participants) | 2 | 5 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (14.14) | 54.5 (15.05) | 49.75 (14.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 1 | 1 | 2
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pathologic Complete Response (pCR)
Description: Pathologic complete response (pCR) defined as the absence of any residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes following completion of neoadjuvant systemic therapy.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | ddACTHP | TCHP
Number analyzed (Participants) | 2 | 5
Participants | 1 | 4

2. Secondary Outcome: Number of Cardiac Toxicity Events
Description: Determination of cardiac toxicity as measured by LVEF, longitudinal strain and troponin.
  Left ventricular ejection fraction (LVEF) measurement of amount of blood being pumped out of the left ventricle of the heart with each contraction.
  Peak systolic longitudinal strain is calculated by averaging the values of peak systolic strain in the basal, mid and apical segments of the LV in 4-, 3- and 2-chamber views on echocardiograms. A value of <-18% or a >15% decline in strain from patient's baseline value will be used as a cut-off value.
  A value of troponin I > 0.08 ng/ml will be considered elevated.
Time Frame: 2 years
Measure: Number; unit: events
Arm/Group | ddACTHP | TCHP
Number analyzed (Participants) | 2 | 5
events | 2 | 2

3. Secondary Outcome: Number of Non-cardiac Toxicities
Description: The frequency of adverse events categorized using CTCAE v4.03
Time Frame: 2 years
Measure: Number; unit: events
Arm/Group | ddACTHP | TCHP
Number analyzed (Participants) | 2 | 5
events | 63 | 120

4. Secondary Outcome: Number of Participants With Breast Conservation
Description: Number of participants with breast-conserving surgery for patients for whom mastectomy was planned before treatment. It would be based on surgical opinion at time of surgery if the tumor was appropriately "downstaged" to perform breast conserving surgery on patients previously recommended to have a mastectomy.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | ddACTHP | TCHP
Number analyzed (Participants) | 2 | 5
Participants | 0 | 0

5. Secondary Outcome: Number of Participants Alive at the End of the Study
Description: Overall Survival - Number of participants alive at the end of the study.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | ddACTHP | TCHP
Number analyzed (Participants) | 2 | 5
Participants | 2 | 5

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | ddACTHP | TCHP
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 2/2 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ddACTHP (N=2) | TCHP (N=5)
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
ALT increase (Hepatobiliary disorders) | 1 | 1
ANC decrease (Blood and lymphatic system disorders) | 1 | 2
Anemia (Blood and lymphatic system disorders) | 2 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 1
AST increase (Hepatobiliary disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 1
chest pain (Cardiac disorders) | 2 | 0
cardiac Troponin-I increase (Cardiac disorders) | 1 | 0
constipation (Gastrointestinal disorders) | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
diarrhea (Gastrointestinal disorders) | 0 | 5
dehydration (Metabolism and nutrition disorders) | 0 | 1
dizziness (Nervous system disorders) | 0 | 1
dry eyes (Eye disorders) | 0 | 1
dry mouth (Gastrointestinal disorders) | 0 | 1
dry skin (Skin and subcutaneous tissue disorders) | 0 | 3
dysgeusia (Nervous system disorders) | 1 | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
edema- limb (General disorders) | 0 | 1
Ejection fraction decrease (Cardiac disorders) | 1 | 0
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
edema-facial (General disorders) | 0 | 1
fatigue (General disorders) | 2 | 4
fever (General disorders) | 0 | 1
Gatro-esophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 1
hot flashes (Vascular disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Lymphocyte count decrease (Blood and lymphatic system disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Parathesia (Nervous system disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2
Platelet count decrease (Blood and lymphatic system disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Skin and subcutaneous tissue disorders other, cysts on groin/pelvis area (Skin and subcutaneous tissue disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Thromboembolic event (Blood and lymphatic system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
WBC decrease (Blood and lymphatic system disorders) | 2 | 3
Watering of eyes (Eye disorders) | 0 | 1
Weight loss (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/78/NCT03329378/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/78/NCT03329378/ICF_001.pdf